CLINICAL TRIAL: NCT00623012
Title: Rapamycin for Prevention of Chronic Graft-Versus-Host Disease
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0702002350
Record Dates: First submitted 2008-02-13; First posted 2008-02-25 (Estimated); Results first posted 2017-02-03 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2016-12

CONDITIONS: Graft Versus Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Sirolimus; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Rapamycin; Drug: Tacrolimus

INTERVENTIONS:
Drug: Rapamycin — Rapamycin will be initiated 24 weeks post SCT, while the patient is on Tacrolimus. The initial dose of rapamycin is 12 mg of loading dose, followed by 4 mg daily. The dose will be adjusted to keep trough level at 3-12 ng/dl. Rapamycin will be continued at the therapeutic dose for 4 additional weeks after Tacrolimus is stopped. Rapamycin will then be tapered off over 2 weeks. The patients will be on 50% of steady state dose for one week and 25% of the steady state dose for the last week.
  Other Names: Sirolimus; Rapamune
Drug: Tacrolimus — Tacrolimus target level is 5-10 ng/dl. Tacrolimus taper will start at 26 weeks post SCT. Tacrolimus will be tapered off over 4-8 weeks. The rate of taper will be 25% every to weeks for patients on 4 mg or more tacrolimus daily. For the patients on 3 mg or less of tacrolimus, the dose will be reduced 1 mg every two weeks, and the last dose will be 1 mg every other day for two weeks.
  Other Names: Prograf

SUMMARY:
The objective of this study is to evaluate feasibility, toxicity and efficacy of using Rapamycin to prevent chronic graft-versus-host-disease (GVHD) during and after the tacrolimus taper in recipients of allogeneic stem cell transplant.

Our hypothesis is that the T cells that can cause chronic GVHD are suppressed but not eliminated by calcineurin inhibitors. Therefore, when the calcineurin inhibitors are discontinued, the T cells may get activated and result in GVHD. Rapamycin on the other hand will allow anergy formation and thus when discontinued, T cells should not get activated. The schedule is designed to have therapeutic rapamycin levels as the tacrolimus is discontinued. Rapamycin will be continued as a single agent for additional 4 weeks and be tapered off in two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Received an allogeneic MSD or MUD PBSCT
* 24 weeks post SCT
* Currently on Tacrolimus for GVHD prophylaxis
* Deemed eligible for tapering off of Tacrolimus by primary BMT physician

Exclusion Criteria:

* Relapsed Disease
* Ongoing GVHD
* Patients whose immunosuppression is being stopped early to treat or prevent relapse
* Patients with pure red cell aplasia due to ABO mismatched donor
* Ongoing thrombotic microangiopathy
* Allergy to rapamycin
* Women of childbearing potential must have a negative serum pregnancy test performed prior to the start of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-02; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Seropian, M.D., Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Population: This is a single arm study:
  Rapamycin: Rapamycin will be initiated 24 weeks post SCT, while the patient is on Tacrolimus. The initial dose of rapamycin is 12 mg of loading dose, followed by 4 mg daily. The dose will be adjusted to keep trough level at 3-12 ng/dl. Rapamycin will be continued at the therapeutic dose for 4 additional weeks after Tacrolimus is stopped. Rapamycin will then be tapered off over 2 weeks. The patients will be on 50% of steady state dose for one week and 25% of the steady state dose for the last week.
  Tacrolimus: Tacrolimus target level is 5-10 ng/dl. Tacrolimus taper will start at 26 weeks post SCT. Tacrolimus will be tapered off over 4-8 weeks. The rate of taper will be 25% every to weeks for patients on 4 mg or more tacrolimus daily. For the patients on 3 mg or less of tacrolimus, the dose will be reduced 1 mg every two weeks, and the last dose will be 1 mg every other day for two weeks.
Period: Overall Study
Arm/Group | Study Population
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Rapamycin Study Arm: Rapamycin: Rapamycin will be initiated 24 weeks post SCT, while the patient is on Tacrolimus. The initial dose of rapamycin is 12 mg of loading dose, followed by 4 mg daily. The dose will be adjusted to keep trough level at 3-12 ng/dl. Rapamycin will be continued at the therapeutic dose for 4 additional weeks after Tacrolimus is stopped. Rapamycin will then be tapered off over 2 weeks. The patients will be on 50% of steady state dose for one week and 25% of the steady state dose for the last week.
  Tacrolimus: Tacrolimus target level is 5-10 ng/dl. Tacrolimus taper will start at 26 weeks post SCT. Tacrolimus will be tapered off over 4-8 weeks. The rate of taper will be 25% every to weeks for patients on 4 mg or more tacrolimus daily. For the patients on 3 mg or less of tacrolimus, the dose will be reduced 1 mg every two weeks, and the last dose will be 1 mg every other day for two weeks.
Arm/Group | Rapamycin Study Arm
Number analyzed (Participants) | 2
Age, Customized [Mean (Full Range); unit: years] | 46 [21 to 70]
Gender [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Improvement of the Rate of Graft Versus Host Disease (GVHD) From the Accepted Rate of 74%.
Description: Percentage of patients free from graft versus host disease
Time Frame: up to 8 weeks
Measure: Number; unit: percentage of patients
Arm/Group | Study Population
Number analyzed (Participants) | 2
percentage of patients | 0

2. Secondary Outcome: Overall Survival
Description: achieved overall survival in regard to leukemia
Time Frame: up to 10 weeks
Measure: Number; unit: participants
Arm/Group | Study Population
Number analyzed (Participants) | 2
participants | 2

3. Secondary Outcome: Disease Free Survival
Description: achieved disease free in regard to leukemia
Time Frame: up to 10 weeks
Measure: Number; unit: participants
Arm/Group | Study Population
Number analyzed (Participants) | 2
participants | 2

ADVERSE EVENTS:
Time Frame: up to 4 months
Description: AE reporting from study entry to one month following completion of study therapy. This period includes study therapy during taper of tacrolimus, continuing for one month after discontinuation of tacrolimus and then a 2 week taper period of study drug. For most subjects this will amount to 3-4 months of monitoring for adverse events.
Groups:
- Study Arm: Rapamycin: Rapamycin will be initiated 24 weeks post SCT, while the patient is on Tacrolimus. The initial dose of rapamycin is 12 mg of loading dose, followed by 4 mg daily. The dose will be adjusted to keep trough level at 3-12 ng/dl. Rapamycin will be continued at the therapeutic dose for 4 additional weeks after Tacrolimus is stopped. Rapamycin will then be tapered off over 2 weeks. The patients will be on 50% of steady state dose for one week and 25% of the steady state dose for the last week.
  Tacrolimus: Tacrolimus target level is 5-10 ng/dl. Tacrolimus taper will start at 26 weeks post SCT. Tacrolimus will be tapered off over 4-8 weeks. The rate of taper will be 25% every to weeks for patients on 4 mg or more tacrolimus daily. For the patients on 3 mg or less of tacrolimus, the dose will be reduced 1 mg every two weeks, and the last dose will be 1 mg every other day for two weeks.
Arm/Group | Study Arm
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
Only 2 patients were enrolled. Early termination of trial, so patients were not followed long enough to see improvement.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No